CLINICAL TRIAL: NCT00099437
Title: A Randomised, Double-Blind, Parallel-group, Multicentre, Phase III Study Comparing the Efficacy and Tolerability of Fulvestrant (FASLODEX™) 500 mg With Fulvestrant (FASLODEX™) 250 mg in Postmenopausal Women With Oestrogen Receptor Positive Advanced Breast Cancer Progressing or Relapsing After Previous Endocrine Therapy
Brief Title: Comparison of Fulvestrant (FASLODEX™) 250 mg and 500 mg in Postmenopausal Women With Oestrogen Receptor Positive Advanced Breast Cancer Progressing or Relapsing After Previous Endocrine Therapy.
Acronym: CONFIRM
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6997C00002; 2004-002371-16 (EudraCT Number)
Record Dates: First submitted 2004-12-13; First posted 2004-12-14 (Estimated); Results first posted 2010-06-15 (Estimated); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: Advanced Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): Fulvestrant 500 mg
  Interventions: Drug: Fulvestrant
- 2 (Experimental): Fulvestrant 250 mg
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: Fulvestrant — intramuscular injection
  Other Names: Faslodex; ZD9238

SUMMARY:
The purpose of this study is to evaluate the efficacy of a new dose of 500 mg Fulvestrant with the standard dose of 250 mg in postmenopausal women with oestrogen receptor positive advanced breast cancer who have failed on a previous endocrine treatment.

ELIGIBILITY:
Inclusion Criteria:

* Breast Cancer has continued to grow after having received treatment with an anti-estrogen hormonal treatment such as tamoxifen or an aromatase inhibitor
* Requiring hormonal treatment
* Postmenopausal women defined as a woman who has stopped having menstrual periods
* Evidence of positive estrogen receptor hormone sensitivity
* Written informed consent to participate in the trial

Exclusion Criteria:

* Treatment with an investigational or non-approved drug within one month
* An existing serious disease, illness, or condition that will prevent participation or compliance with study procedures
* A history of allergies to any active or inactive ingredients of Faslodex (i.e. castor oil)
* Treatment with more than one regimen of chemotherapy for advanced breast cancer
* Treatment with more than one regimen of hormonal treatment for advanced breast cancer

Ages: 45 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 736 (Actual)
Dates: Start 2005-02-13 (Actual); Primary Completion 2009-02-27 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Faslodex Medical Science Director, MD, Study Director — AstraZeneca
Locations (93):
- United States (14):
  - Research Site, Casa Grande, Arizona
  - Research Site, Fountain Valley, California
  - Research Site, New Britain, Connecticut
  - Research Site, Crystal River, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Urbana, Illinois
  - Research Site, Rosedale, Maryland
  - Research Site, Detroit, Michigan
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Voorhees Township, New Jersey
  - Research Site, Greenville, North Carolina
  - Research Site, Pasadena, Texas
  - Research Site, West Bend, Wisconsin
- Belgium (7):
  - Research Site, Brasschaat
  - Research Site, Brussels
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Hasselt
  - Research Site, Liège
  - Research Site, Turnhout
- Brazil (6):
  - Research Site, Barretos
  - Research Site, Londrina
  - Research Site, Porto Alegre
  - Research Site, Recife
  - Research Site, Salvador
  - Research Site, São Paulo
- Chile (2):
  - Research Site, Antofagasta
  - Research Site, Santiago
- Colombia (2):
  - Research Site, Bogotá
  - Research Site, Cali
- Czechia (6):
  - Research Site, Brno
  - Research Site, České Budějovice
  - Research Site, Pardubice
  - Research Site, Prague
  - Research Site, Tábor
  - Research Site, V Uvalu 84
- Hungary (3):
  - Research Site, Nyíregyháza
  - Research Site, Székesfehérvár
  - Research Site, Szombathely
- India (11):
  - Research Site, Ansārinagar
  - Research Site, Bhopal
  - Research Site, Hyderabad
  - Research Site, Jaipur
  - Research Site, Kolkata
  - Research Site, Manipal
  - Research Site, Marg Jaipur
  - Research Site, Mumbai
  - Research Site, Pune
  - Research Site, Trivandrum
  - Research Site, Vellore
- Italy (7):
  - Research Site, Aviano
  - Research Site, Bergamo
  - Research Site, Carpi
  - Research Site, Genova
  - Research Site, Prato
  - Research Site, Reggio Emilia
  - Research Site, Varese
- Research Site, Floriana, Malta
- Mexico (2):
  - Research Site, Mexico City
  - Research Site, México
- Poland (3):
  - Research Site, Bialystok
  - Research Site, Lodz
  - Research Site, Poznan
- Russia (10):
  - Research Site, Ivanovo
  - Research Site, Kazan, Tatarstan
  - Research Site, Krasnodar
  - Research Site, Lipetsk
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Obninsk
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Yaroslavl
- Slovakia (4):
  - Research Site, Bardejov
  - Research Site, Bratislava
  - Research Site, Nitra
  - Research Site, Trnava
- Spain (6):
  - Research Site, A Coruña
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Oviedo
  - Research Site, Salamanca
  - Research Site, Seville
- Ukraine (8):
  - Research Site, Cherkasy
  - Research Site, Dnipro
  - Research Site, Donetsk
  - Research Site, Kyiv
  - Research Site, Lviv
  - Research Site, Sumy
  - Research Site, Ternopil
  - Research Site, Uzhhorod
- Research Site, Caracas, Venezuela

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Wedam SB, Beaver JA, Amiri-Kordestani L, Bloomquist E, Tang S, Goldberg KB, Sridhara R, Ibrahim A, Kim G, Kluetz P, McKee A, Pazdur R. US Food and Drug Administration Pooled Analysis to Assess the Impact of Bone-Only Metastatic Breast Cancer on Clinical Trial Outcomes and Radiographic Assessments. J Clin Oncol. 2018 Apr 20;36(12):1225-1231. doi: 10.1200/JCO.2017.74.6917. Epub 2018 Mar 9. PMID 29522361
- See also: CSP-D6997C00002.PDF — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=589&filename=CSP-D6997C00002.PDF
- See also: D6997C00002 Study Report Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=589&filename=CSR-D6997C00002.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Fulvestrant 250 mg: Fulvestrant 250 mg Intramuscular Injection every 28 days
- Fulvestrant 500 mg: Fulvestrant 500 mg Intramuscular Injection every 28 days plus 500 mg on day 14
Period: Overall Study
Arm/Group | Fulvestrant 250 mg | Fulvestrant 500 mg
Started | 374 (randomised patients) | 362 (randomised patients)
Completed | 8 (ongoing study treatment at survival follow-up data cut-off) | 13 (ongoing study treatment at survival follow-up data cut-off)
Not Completed | 366 | 349
Not completed — Lost to Follow-up | 30 | 33
Not completed — Death | 293 | 261
Not completed — Withdrawal by Subject | 6 | 10
Not completed — Ongoing in FU but not on treatment | 37 | 45

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fulvestrant 250 mg | Fulvestrant 500 mg | Total
Number analyzed (Participants) | 374 | 362 | 736
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.8 (11.94) | 61.0 (11.47) | 60.9 (11.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 374 | 362 | 736
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression (TTP)
Description: Median time (in months) from randomisation until objective disease progression or death (in the absence of objective progression).
Time Frame: RECIST(Response Evaluation Criteria in Solid Tumors ) tumour assessments carried out every 12 weeks (+/- 2 weeks) from randomisation for study duration (48 months)
Measure: Median (Full Range); unit: months
Arm/Group | Fulvestrant 250 mg | Fulvestrant 500 mg
Number analyzed (Participants) | 374 | 362
months | 5.5 [0 to NA] — Not Applicable - not all participants had an event at time of analysis, max time censored | 6.5 [0 to NA] — Not Applicable - not all participants had an event at time of analysis, max time censored

2. Secondary Outcome: Objective Response Rate (ORR)
Description: Using the RECIST scan data, an objective response (OR) is defined as a patient having a best overall response of either complete response (CR) or partial response (PR) which is subsequently confirmed as per RECIST. ORR is defined as the percentage of patients with OR.
Time Frame: RECIST tumour assessments carried out every 12 weeks (+/- 2 weeks) from randomisation for study duration (48 months)
Population: All patients with measurable disease at baseline.
Measure: Number; unit: Percentage of patients
Arm/Group | Fulvestrant 250 mg | Fulvestrant 500 mg
Number analyzed (Participants) | 261 | 240
Percentage of patients | 14.6 | 13.8

3. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: A Clinical Benefit (CB) responder is defined as a patient having a best overall response of CR, PR or SD (stable disease) >=24 weeks. The Clinical Benefit Rate is the percentage of patients with CB.
Time Frame: Clinical Benefit from the sequence of RECIST scan data for study duration (48 months) . RECIST (Response Evaluation Criteria in Solid Tumours) scans were performed every 12 weeks (+/- 2 weeks) from randomisation for study duration (48 months)
Measure: Number; unit: Percentage of patients
Arm/Group | Fulvestrant 250 mg | Fulvestrant 500 mg
Number analyzed (Participants) | 374 | 362
Percentage of patients | 39.6 | 45.6

4. Secondary Outcome: Duration of Response (DoR)
Description: Time from randomisation until objective progression or death (in the absence of objective progression), measured only in those patients who achieve a confirmed complete response (CR) or confirmed partial response (PR)
Time Frame: RECIST tumour assessments carried out every 12 weeks (+/- 2 weeks) from randomisation for study duration (48 months)
Measure: Median (Full Range); unit: Time (in months)
Arm/Group | Fulvestrant 250 mg | Fulvestrant 500 mg
Number analyzed (Participants) | 38 | 33
Time (in months) | 16.4 [3.7 to NA] — Not Applicable - not all participants had an event at time of analysis, max time censored | 19.4 [5.7 to NA] — Not Applicable - not all participants had an event at time of analysis, max time censored

5. Secondary Outcome: Duration of Clinical Benefit (DoCB)
Description: Time from randomisation until objective progression or death (in the absence of objective progression), measured only in those patients who achieve a confirmed complete response (CR), confirmed partial response (PR), or stable disease (SD) >=24 weeks
Time Frame: RECIST tumour assessments carried out every 12 weeks (+/- 2 weeks) from randomisation for study duration (48 months)
Measure: Median (Full Range); unit: Time (in months)
Arm/Group | Fulvestrant 250 mg | Fulvestrant 500 mg
Number analyzed (Participants) | 148 | 165
Time (in months) | 13.9 [3.7 to NA] — Not Applicable - not all participants had an event at time of analysis, max time censored | 16.6 [2.5 to NA] — Not Applicable - not all participants had an event at time of analysis, max time censored

6. Secondary Outcome: Overall Survival (OS)
Description: Median time (in months) from randomisation until death (from any cause) (analysis at 50% deaths )
Time Frame: Overall Survival is equivalent to time to death. For this endpoint, all deaths occurring for study duration (48 months)
Population: All patients with measurable disease at baseline.
Measure: Median (Full Range); unit: Time (in months)
Arm/Group | Fulvestrant 250 mg | Fulvestrant 500 mg
Number analyzed (Participants) | 374 | 362
Time (in months) | 22.8 [0.2 to NA] — Not Applicable - not all participants had an event at time of analysis, max time censored | 25.1 [0.1 to NA] — Not Applicable - not all participants had an event at time of analysis, max time censored

7. Secondary Outcome: Change From Randomisation in Trial Outcome Index (TOI) Over the Course of the Study
Description: Mean (and standard deviation) change from randomisation until treatment discontinuation in TOI (defined as the first visit response of 'worsened' which is a decrease in TOI from baseline of 5 points or more) using the Kaplan-Meier method. If a subject has not shown a reduction of 5 points or more at the time of analysis then the observation will be right censored using the last QOL assessment date. Trial Outcome Index (TOI) is derived from the FACT-B questionnaire (Cella et al, 1993) by adding together the scores from the following 3 subscales; Physical well-being (PWB), Functional well-being (FWB) and Breast cancer subscale (BCS). The TOI score range is 0-92 with the higher scores representing the more favourable outcomes. Data were collected from a subgroup of patients.
Time Frame: TOI questionnaires were completed every 4 weeks from randomisation until week 24 and then again at treatment discontinuation, for study duration (48 months)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Fulvestrant 250 mg | Fulvestrant 500 mg
Number analyzed (Participants) | 35 | 34
Scores on a scale | -5.9 (9.89) | -7.5 (13.72)

8. Secondary Outcome: Overall Survival (OS) - Follow-up
Description: Overall Survival is equivalent to time to death. For this endpoint, all deaths occurring during the study as a whole until the data cut-off for the survival extension (31st October 2011) are presented (analysis at 75% deaths)
Time Frame: Median time (in months) from randomisation until death (from any cause),up to 80 months
Population: All randomised patients
Measure: Median (Full Range); unit: months
Arm/Group | Fulvestrant 250 mg | Fulvestrant 500 mg
Number analyzed (Participants) | 374 | 362
months | 22.3 [0.2 to NA] — Not Applicable - not all participants had an event at time of analysis, max time censored | 26.4 [0.1 to NA] — Not Applicable - not all participants had an event at time of analysis, max time censored

ADVERSE EVENTS:
Time Frame: SAE- From baseline up to October 31st 2011; AE- From baseline up to 28th February 2009
Description: 1 participant was randomised to fulvestrant 500 mg but did not receive any treatment. AEs have been collected up to primary data cut off. SAEs have been collected up to follow-up phase data cut-off.
Arm/Group | Fulvestrant 250 mg | Fulvestrant 500 mg
Serious Adverse Events (participants affected / at risk) | 27/374 | 35/361
Other Adverse Events (participants affected / at risk) | 235/374 | 241/361
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fulvestrant 250 mg (N=374) | Fulvestrant 500 mg (N=361)
Anaemia (Blood and lymphatic system disorders) | 1 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Cardiopulmonary Failure (Cardiac disorders) | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 2 | 0
Myocardial Ischaemia (Cardiac disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Duodenal Ulcer Perforation (Gastrointestinal disorders) | 0 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Adverse Drug Reaction (General disorders) | 0 | 1
Death (General disorders) | 0 | 1
General Physical Health Deterioration (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 2
Bronchopneumonia (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 0 | 2
Urinary Tract Infection (Infections and infestations) | 0 | 1
Viral Infection (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1
Contrast Media Reaction (Injury, poisoning and procedural complications) | 0 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 2 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 1
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 | 0
Head Injury (Injury, poisoning and procedural complications) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Benign Mediastinal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intestinal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral Ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 0 | 1
Meningorrhagia (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Completed Suicide (Psychiatric disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
Venous Thrombosis Limb (Vascular disorders) | 0 | 1
Arterial Thrombosis Limb (Vascular disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
Iliac Artery Embolism (Vascular disorders) | 1 | 0
Venous Thrombosis (Vascular disorders) | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 1
ASTHENIA (General disorders) | 0 | 1
INFECTIOUS PERITONITIS (Infections and infestations) | 0 | 1
FALL (Injury, poisoning and procedural complications) | 1 | 0
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fulvestrant 250 mg (N=374) | Fulvestrant 500 mg (N=361)
Nausea (Gastrointestinal disorders) | 51 | 35
Vomiting (Gastrointestinal disorders) | 20 | 21
Injection Site Pain (Gastrointestinal disorders) | 34 | 42
Fatigue (Gastrointestinal disorders) | 24 | 27
Asthenia (Gastrointestinal disorders) | 23 | 21
Anorexia (Metabolism and nutrition disorders) | 14 | 22
Back Pain (Musculoskeletal and connective tissue disorders) | 40 | 26
Bone Pain (Musculoskeletal and connective tissue disorders) | 28 | 34
Arthralgia (Musculoskeletal and connective tissue disorders) | 29 | 29
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 26 | 25
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 12 | 20
Headache (Nervous system disorders) | 25 | 28
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 19
Hot Flush (Vascular disorders) | 22 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that they cannot publish any information to do with the trial without written consent from Quintiles.